CLINICAL TRIAL: NCT05710484
Title: Investigating the Impact of Inferior Alveolar Nerve Block Anesthesia on Acoustic Voice Quality Using a Within-subject Design
Brief Title: Voice Quality Changes With IANB Anesthesia
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Other Study IDs: MUDHF_FB_003
Record Dates: First submitted 2023-01-25; First posted 2023-02-02 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia, Local; Voice Change
Keywords: Voice Quality; Anesthesia, Dental; Mandibular Nerve; Lingual Nerve; Speech Acoustics
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inferior alveolar nerve block anesthesia cohort: This group will consist of participants who are undergoing procedures that require mandibular anesthesia as routine part of care. Participants in this group will have voice recordings taken before and after the administration of anesthesia. The aim is to assess any changes in voice characteristics attributable to the effect of the anesthesia.

SUMMARY:
Background: Inferior alveolar nerve block anesthesia is commonly used in dental procedures, but its effect on the voice quality is not well understood. The aim of this study is to investigate the effect of mandibular anesthesia on the acoustic voice quality index.

Objective: The primary objective of this study is to determine the effect of mandibular anesthesia on the acoustic voice quality index.

Design: This is a within-subject study design. Participants will be recruited from a local dental clinic and will be adults aged 18 years or older. The participants will have the acoustic voice quality index measured before and after the administration of mandibular anesthesia. The parameters that will be measured include acoustic voice quality index and self ........ The data will be analyzed using appropriate statistical techniques.

Expected Outcome: The study is expected to provide insights into the effect of mandibular anesthesia on the acoustic voice quality index. The results of this study may help in understanding the impact of mandibular anesthesia on voice quality and may have implications for dental practitioners and patients who receive mandibular anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* able to communicate in the local language
* no history of voice disorders or speech therapy
* no history of any diseases or conditions that could affect voice quality.

Exclusion Criteria:

* pregnant or breastfeeding women
* individuals with a history of allergies or adverse reactions to anesthesia
* individuals with a history of any diseases or conditions that could affect voice quality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults aged 18 years or older who are scheduled to receive inferior alveolar nerve block anesthesia as part of their dental procedure.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Acoustic Voice Analyze measurements; Motor Speech Profile (MSP) | Immediate before inferior alveolar nerve block anesthesia, immediately after inferior alveolar nerve block anesthesia roughly 5 minutes later
  Motor Speech Profile (MSP), is being used for accuracy and straightness of motor performance of speech. An inaccurate, inconsistent or abnormal oral-diadochokinetic performance may indicate disturbances in central nervous system or peripheral sensory motor functions. The software based on different protocols that provide different motor speech patterns such as oral diadochokinetic (DDK) rate, second formant transition rate, and syllable rate.
Change in Acoustic Voice Analyze measurements; Multi-dimensional voice program (MDVP) | Immediate before inferior alveolar nerve block anesthesia, immediately after inferior alveolar nerve block anesthesia roughly 5 minutes later
  Multi-dimensional voice program (MDVP), basically, it is a computer program which analyzes various aspects of voice. It can provide many of acoustic parameters from a voice sample. It is based on a continuous vowel: /a/.
Change in Acoustic Voice Analyze measurements; Analysis of dysphonia in speech and voice (ADSV) | Immediate before inferior alveolar nerve block anesthesia, immediately after inferior alveolar nerve block anesthesia roughly 5 minutes later
  Analysis of dysphonia in speech and voice (ADSV), evaluates frequency domain parameters. It is based on 2 different vowels ((/a/ and /i/) from Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) and 6 different sentences. Every single sentence provides different voice analyses such as, containing all the vowels, making sounds with or without glottal attack, nasal sounds or explosive sounds.
Change in Acoustic Voice Analyze measurements;Acoustic Voice Quality Index (AVQI) | Immediate before inferior alveolar nerve block anesthesia, immediately after inferior alveolar nerve block anesthesia roughly 5 minutes later
  Acoustic Voice Quality Index (AVQI), measures the perceived quality of a voice signal. It is based on evaluating several acoustic parameters that are known to be related to the perceived quality of speech. These parameters include measures of loudness, pitch and spectral tilt as well as measures of the presence of noise and other distortions in the signal.

SECONDARY OUTCOMES:
Change in BORG Scale (CR-10) | Exercise timing is immediate before inferior alveolar nerve block anesthesia, holding a dental mirror with only lips and tongue, for 2 minutes
  A method for rating perceived effort and the CR-10 is a "semi-public/semi-public" tool for different boundaries and different measured structures. It is required for participants to correctly score the perceived effort against the variable during the experimental procedure. An exercise can be planned for setting the extreme points of the experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barsties V Latoszek B, Ulozaite-Staniene N, Petrauskas T, Uloza V, Maryn Y. Diagnostic Accuracy of Dysphonia Classification of DSI and AVQI. Laryngoscope. 2019 Mar;129(3):692-698. doi: 10.1002/lary.27350. Epub 2018 Sep 10. PMID 30203473
- [Background] Corbett IP, Kanaa MD, Whitworth JM, Meechan JG. Articaine infiltration for anesthesia of mandibular first molars. J Endod. 2008 May;34(5):514-8. doi: 10.1016/j.joen.2008.02.042. PMID 18436027
- [Background] Correia JM, Caballero-Gaudes C, Guediche S, Carreiras M. Phonatory and articulatory representations of speech production in cortical and subcortical fMRI responses. Sci Rep. 2020 Mar 11;10(1):4529. doi: 10.1038/s41598-020-61435-y. PMID 32161310
- [Background] Hogikyan ND, Sethuraman G. Validation of an instrument to measure voice-related quality of life (V-RQOL). J Voice. 1999 Dec;13(4):557-69. doi: 10.1016/s0892-1997(99)80010-1. PMID 10622521
- [Background] Maryn Y, Corthals P, Van Cauwenberge P, Roy N, De Bodt M. Toward improved ecological validity in the acoustic measurement of overall voice quality: combining continuous speech and sustained vowels. J Voice. 2010 Sep;24(5):540-55. doi: 10.1016/j.jvoice.2008.12.014. Epub 2009 Nov 2. PMID 19883993
- [Background] Nanjundeswaran C, Jacobson BH, Gartner-Schmidt J, Verdolini Abbott K. Vocal Fatigue Index (VFI): Development and Validation. J Voice. 2015 Jul;29(4):433-40. doi: 10.1016/j.jvoice.2014.09.012. Epub 2015 Mar 17. PMID 25795356
- [Background] Sirin S, Ogut MF, Bilgen C. Reliability and validity of the Turkish version of the Vocal Fatigue Index. Turk J Med Sci. 2020 Jun 23;50(4):902-909. doi: 10.3906/sag-1908-105. PMID 32421276
- [Background] Yesilli-Puzella G, Tadihan-Ozkan E, Maryn Y. Validation and Test-Retest Reliability of Acoustic Voice Quality Index Version 02.06 in the Turkish Language. J Voice. 2022 Sep;36(5):736.e25-736.e32. doi: 10.1016/j.jvoice.2020.08.021. Epub 2020 Sep 20. PMID 32962941
- [Derived] Sahin C, Bayram F, Yilmaz G, Gocmen GB, Konrot A. Effect of inferior alveolar and lingual nerve block anesthesia on acoustic voice quality and speech effort: A within-subject study. J Am Dent Assoc. 2025 Dec;156(12):982-990. doi: 10.1016/j.adaj.2025.08.021. Epub 2025 Oct 14. PMID 41085515